CLINICAL TRIAL: NCT06723093
Title: Impact of a Social Medicine Housing Program on the Health and Healthcare Utilization of Adults Who Are Unhoused and Have Complex Health Needs
Brief Title: Evaluation of a Supportive Housing Program for Adults Who Are Unhoused and Have Complex Health Needs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Andrew Boozary, Executive Director, Population Health and Social Medicine Gattuso Centre for Social Medicine, University Health Network, University Health Network, Toronto
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-5519
Record Dates: First submitted 2024-11-21; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Homeless Persons
Keywords: homelessness

STUDY DESIGN:
Intervention Model Description: The study design is a cohort study with a propensity score-matched control group and difference-in-difference analysis to evaluate intervention effectiveness. A hybrid type 1 effectiveness-implementation study framework is used that incorporates mixed methods to determine clinical effectiveness and explore implementation and participant well-being.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- University Health Network Standard Care (Experimental): The Social Medicine Housing Initiative is part of standard care and is not contingent on participating in any research activities. Patients who participate in the Housing Initiative will have the option to participate in the research study.
  The Social Medicine Housing Initiative provides a housing-first approach which offers housing to individuals without prerequisites (e.g., requiring cessation of substance use, adherence to treatment). Through the Initiative, patients will receive access to permanent supportive housing and support services based on the Social Medicine model. Participants will not only have access to housing but will also be provided with customized social and medical support within and beyond the University Health Network, tailored to their specific needs and preferences.
  Interventions: Behavioral: Social Medicine Housing Initiative
- Propensity score matched cohort (No Intervention): The Institute of Clinical Evaluative Sciences of Canada database will provide health administrative data on the Housing Initiative individuals and similar individuals. Each individual in the treatment arm will be matched with four individuals (1:4 pair) in the control arm who are observationally similar. The propensity score-matched cohort method will control for demand-side characteristics that reflect the utilization of health care services, focusing on the use of emergency department visits and inpatient hospital days, nursing home use, and inpatient utilization for severe mental illness. To assess whether the propensity score model has adequately specified, the authors will examine whether the distribution of measured baseline covariates is similar between treated and untreated subjects with the same estimated propensity score.

INTERVENTIONS:
Behavioral: Social Medicine Housing Initiative — Through the Social Medicine Housing Initiative, patients will receive access to permanent supportive housing and support services based on a social medicine model. The Housing Initiative provides a housing-first approach which offers housing to individuals without prerequisites (e.g., requiring cessation of substance use, adherence to treatment). Housing will be provided through a rent-geared-to-income model, with participants paying up to 30 percent of their income towards rent.
  Participants will also be provided with customized social and medical support within and beyond the University Health Network, tailored to their specific needs and preferences. Patient care will be a collaborative effort involving the housing provider, the Social Medicine team, and community agencies.
  Arms: University Health Network Standard Care

SUMMARY:
The study design is a cohort study with a propensity score-matched control group and difference-in-difference analysis to evaluate intervention effectiveness. A hybrid type 1 effectiveness-implementation study framework is used that incorporates mixed methods to determine clinical effectiveness and explore implementation and participant well-being. Participants are selected based on their utilization of health services. Selection favoured those individuals with the most health service utilization. A control group will be created by selecting individuals from administrative hospital records that are propensity-score matched to the individuals in the treatment group (1:4 pair). The hybrid type 1 effectiveness-implementation study framework was used to guide the selection of study aims and outcomes to focus primarily on clinical effectiveness, while also exploring implementation-related factors. The primary objective of the study is to evaluate the impact of the Initiative on the number of emergency department visits and days spent in the hospital. The secondary objectives are to 2) evaluate the impact of the Initiative on program participants' health and well-being, 3) evaluate the implementation of the Initiative and assess program fidelity and barriers, and 4) to calculate the cost avoidance and cost-effectiveness of the Initiative.

DETAILED DESCRIPTION:
The study design is a cohort study with a propensity score-matched control group and difference-in-difference analysis to evaluate intervention effectiveness. A hybrid type 1 effectiveness-implementation study framework is used that incorporates mixed methods to determine clinical effectiveness and explore implementation and participant well-being.

Using a quasi-experimental design approach, participants are not randomly assigned to the intervention group. Participants are selected based on their utilization of health services, satisfying the other inclusion criteria, and accepting to participate in the Initiative. Selection favored those individuals with the most health service utilization. All intervention participants will be invited to participate in the evaluation study. A control group will be created by selecting individuals from administrative hospital records that are propensity score matched to the individuals in the treatment group. Four control individuals will be selected for every one treatment individual (1:4 pair). Patient data from multiple time points, before and after intervention implementation, will be used to strengthen the analysis and to compare immediate and longer-term effects to the treatment group. The propensity-score matching procedure is described below.

The hybrid type 1 effectiveness-implementation study framework was used to guide the selection of study aims and outcomes to focus primarily on clinical effectiveness, while also exploring implementation-related factors. This approach helps to combine questions concerning the effectiveness of the intervention with questions about how best to implement it. The clinical, service, and implementation outcomes, according to Proctor's Outcomes for Implementation Research, will be analyzed in conjunction to provide a complete understanding of the program mechanisms of change.

Mixed methods will be used to combine quantitative and qualitative data in a convergent approach. The quantitative and qualitative data will be collected in parallel, primarily, to merge the information and compare the results for triangulation of the findings. Triangulating data from multiple methods and sources will allow us to comprehensively answer the evaluation questions, minimize bias, and increase the credibility of the results. Data collection sources are described below.

All participants that were selected and agreed to participate in the Social Medicine Housing Initiative will be invited to participate in the study. The tenants of Social Medicine Housing Initiative must consent to participate in the study. The participants will be housed at the newly constructed housing building in Toronto or will be housed in units that become available throughout the city. There are no exclusion criteria that would exclude participants who are receiving housing from participating in the research study. If participants are able to independently provide consent, or do not want to provide consent for the study, they will be excluded.

To qualify to participate in the Social Medicine Housing Initiative, patients must have had 2 or more inpatient admissions or 6 or more visits to the emergency department in the past 6 months. They must also be currently without housing, which is defined as having spent at least one night in a shelter or having received assistance from city-funded street outreach providers in the past 90 days. Alternatively, the patient can participate in Social Medicine Housing Initiative if they identify as Indigenous. Historically marginalized groups, including people with disabilities, women, gender-diverse individuals, and Indigenous people, are given priority for housing.

University Health Network program coordinators will identify potential participants of the Social Medicine Housing Initiative through the health system data of the University Health Network hospitals. Once identified, the potential participant will be asked by a member of the community organization that will manage the housing (Fred Victor Organization) if they would like to move into the housing and participate in the Social Medicine Housing Initiative. After the participants confirm their involvement in the Social Medicine Housing Initiative, coordinators at the University Health Network will speak with them to invite them to participate in the study and to conduct the informed consent process. University Health Network coordinators will explain the purpose, process, risks and benefits of the study. Participants will then confirm their enrollment in the study by providing written informed consent.

All tenant study participants will be asked to participate in mixed-methods surveys and in-depth interviews to assess their well-being, their perception of the program, and their personal journey. All interviews will last between 45 and 60 minutes and will be audio-recorded so they can be transcribed for analysis. All surveys will be conducted in the housing facility or another private location that is comfortable for the participant. The surveys will be administered through the REDcap application for managing online surveys and databases(8). The survey will be conducted by a member of the University Health Network research team using a smartphone or tablet. University Health Network will hire research and interview specialists with experience in mixed-methods surveys and experience working with vulnerable populations.

Administrative health data will be obtained through an Applied Health Research Questions Research Project from the Institute of Clinical Evaluative Sciences of Canada. ICES is a non-profit, independent research instate funding by the Ontario Ministry of Health and the Ministry of Long-Term Care. The Institute of Clinical Evaluative Sciences of Canada has legal status under Ontario's health information privacy law which allows it to collect and analyze healthcare and demographic data, without consent, for health system evaluation and improvement. Using a data sharing agreement, an The Institute of Clinical Evaluative Sciences of Canada researcher will provide relevant information on health care resource utilization for study participants. The administrative health data housed at the Institute of Clinical Evaluative Sciences of Canada will be used to conduct the propensity score matching and to obtain the data to assess the outcomes described in Aim 1, Aim 2, and Aim 4. The Institute of Clinical Evaluative Sciences of Canada data will be used to measure the following indicators: Emergency department visits, Days spent in the hospital, Inpatient Utilization for Substance Use Disorder, Inpatient Utilization for Severe Mental Illness, Mortality, Primary Care Visits, Specialist Visits.

ELIGIBILITY:
Inclusion Criteria:

* The Housing Initiative is part of standard care and is not contingent on participating in any research activities. Patients that participate in the Housing Initiative will have the option to participate in the research study.
* To qualify for housing through the initiative, patients must have had 2 or more inpatient admissions or 6 or more visits to the emergency department in the past 6 months. They must also either identify as Indigenous or be currently without housing, which is defined as having spent at least one night in a shelter or having received assistance from city-funded street outreach providers in the past 90 days. Historically marginalized groups, including people with disabilities, women, gender-diverse individuals, and Indigenous people, are given priority for housing. Eligible patients are prioritized for housing offers based on their use of the University Health Network emergency departments in the past year.

There are no exclusion criteria that would disqualify participants from participating in the research study if they have already enrolled in the Social Medicine Housing Initiative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of emergency department visits | 30 Months
  The primary objective of the study is to evaluate the impact of the Social Medicine Housing Initiative on the number of emergency department visits for University Health Network super utilizers compared to a propensity score-matched cohort. It is hypothesized that study participants who participate in the Housing Initiative will show a reduction in acute care utilization (emergency department visits) during the 30-month outcome ascertainment period.
Days spent in the hospital | 30 Months
  The primary objective of the study is to evaluate the impact of the Social Medicine Housing Initiative on the number of days spent in the hospital for UHN super-utilizers compared to a propensity score-matched cohort. It is hypothesized that study participants who participate in the Housing Initiative will show a reduction in acute care utilization (in-patient hospital days) during the 30-month outcome ascertainment period

SECONDARY OUTCOMES:
Tenant Health status | 30 months
  A "Tenant Well-being Survey" was created using validated scales from the Massachusetts Behavioral Risk Factor Surveillance (BRFSS) questionnaires. The Well-being Survey will first be administered to the study participants at baseline and again at (approximately) month 8, month 16, month 30, and if/when a participant chooses to leave the program.
  The "Tenant Well-being Survey" will include 10 self-reported questions related to the health of tenants, including perceived access to health care, number of days their health was not good in the past month, barriers to accessing health care ( e.g. transportation, cost appointment scheduling), and preferred location to accessing health care services). Scores will not be aggregated for the health care measures.
Tenant Mental health | 30 months
  A "Tenant Well-being Survey" was created using validated scales from the Massachusetts Behavioral Risk Factor Surveillance (BRFSS) questionnaires. The Well-being Survey will first be administered to the study participants at baseline and again at (approximately) month 8, month 16, month 30, and if/when a participant chooses to leave the program.
  The "Tenant Well-being Survey" will include 9 self-reported questions related to the mental health of tenants, including: a scale of how many days they felt anxious in the past 30 days, a scale of how many days they felt depressed in the past 30 days, if they have received professional counselling for their mental health, barriers to accessing mental health care ( e.g. transportation, cost appointment scheduling), and perceived access to informal support systems. Scores will not be aggregated for the mental health care measures.
Tenant Substance Use | 30 months
  A "Tenant Well-being Survey" was created using validated scales from the Massachusetts Behavioral Risk Factor Surveillance (BRFSS) questionnaires. The Well-being Survey will first be administered to the study participants at baseline and again at (approximately) month 8, month 16, month 30, and if/when a participant chooses to leave the program.
  The "Tenant Well-being Survey" will include 7 self-reported questions related to the substance use, including: number of drinks in the past 30 days, number of overdoses in the past 30 days, impact of substance use on important activities, and use despite negative consequences. Scores will not be aggregated for the mental health care measures.
Tenant history of violence | 30 months
  A "Tenant Well-being Survey" was created using validated scales from the Massachusetts Behavioral Risk Factor Surveillance (BRFSS) questionnaires. The Well-being Survey will first be administered to the study participants at baseline and again at (approximately) month 8, month 16, month 30, and if/when a participant chooses to leave the program.
  The "Tenant Well-being Survey" will include 2 self-reported questions related to experiences of violence in the last 6 months and 1 self-reported question on history of sexual violence in the last 6 months.

OTHER OUTCOMES:
Health care expenditure analysis | 30 months
  The study aims to look at the impact of the program on those that receive the resources from the program, to determine if the cost of the program is justifiable considering the reduction in healthcare utilization. Cost data will be obtained from the Institute of Clinical Evaluative Sciences of Canada (ICES) on hospital health service cost reports. These databases can also be used to estimate healthcare costs for health services covered by the government using validated individual-level costing algorithms that combine the frequency and intensity of resource utilization with a weighted per unit cost. It is hypothesized that the Initiative will reduce the cost-burden incurred by the health system from serving the study participants.
Cost effectiveness analysis | 30 months
  The study aims to look at the impact of the program on those that receive the resources from the program, to determine if the cost of the program is justifiable considering the reduction in healthcare utilization. Cost data will be obtained from the Institute of Clinical Evaluative Sciences of Canada (ICES) on hospital health service cost reports. These databases can also be used to estimate healthcare costs for health services covered by the government using validated individual-level costing algorithms that combine the frequency and intensity of resource utilization with a weighted per unit cost. A cost-effectiveness analysis will be conducted based on the costs of the Initiative compared to cost avoidance within the health care system. It is hypothesized that the cost of providing the Initiative will be less than the cost-saved from the reduced health system utilization created by it.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Boozary, MD MPP CCFP, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - University Health Network, Toronto, Ontario
  - 90 Dunn, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No